CLINICAL TRIAL: NCT03585712
Title: A Prospective, Multi-center, Randomized, Cross-over Study to Assess the Effect of Norgestrel 75 mcg on Cervical Mucus and Ovarian Activity During Perfect Use, After One Delayed Intake and After a Missed Pill
Brief Title: Effect of Norgestrel 75 mcg on Cervical Mucus and Ovarian Activity During Perfect Use, After One Delayed Intake and After a Missed Pill
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HRA Pharma (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 151042-002
Record Dates: First submitted 2018-07-05; First posted 2018-07-13 (Actual); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Contraception
Keywords: Birth Control; Progestin Only Pill; Estrogen Free Pill; Norgestrel; Oral Contraception; Female Contraception; Cervical Mucus; Ovarian Activity
MeSH Terms: interventions — Norgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Delayed then Missed Pill (Other): Treatment period 2, Day 42 +/- 3 days: 6 hour delayed intake of Norgestrel 75 mcg Treatment period 3, Day 70 +/- 3 days: missed pill of Norgestrel 75 mcg
  Interventions: Drug: Norgestrel 0.075 mg
- Arm B: Missed then Delayed Pill (Other): Treatment period 2, Day 42 +/- 3 days: missed pill of Norgestrel 75 mcg Treatment period 3, Day 70 +/- 3 days: 6 hour delayed intake of the pill of Norgestrel 75 mcg
  Interventions: Drug: Norgestrel 0.075 mg

INTERVENTIONS:
Drug: Norgestrel 0.075 mg — Subjects will take norgestrel 75 mcg every day at the same time for three 28-day treatment periods, except for 1 specific day during treatment period 2 and treatment period 3
  Other Names: Norgestrel 75 mcg

SUMMARY:
Norgestrel 75 mcg is a progestin-only pill (POP), which is a kind of oral birth control pill.

To be effective in preventing pregnancy, this kind of birth control pill is supposed to be taken every day at the same time, without delaying the intake for more than 3 hours.

This study aims to find out if taking the pill 6 hours late or not taking it for one day will affect the way it works.

DETAILED DESCRIPTION:
This study is an exploratory, prospective, multi-center, randomized, cross-over study to assess the effect of norgestrel 75 mcg on cervical mucus and ovarian activity during reported perfect daily use, after a delayed intake of 6 hours and after a missed pill.

After a screening period up to one month, depending on the menstrual cycle of the subject, the subjects will take norgestrel 75 mcg for three 28-day treatment periods, every day at the same time except for one day in the middle of treatment period 2 and treatment period 3 where they will either take it 6 hours late or not take it.

In week 5 (1st visit of treatment period 2), they will be randomized to 2 sequences, either 6 hours delayed intake in treatment period 2 and missed pill in treatment period 3 or the opposite.

After the end of treatment period 3, a follow-up up to 12 days may be required to follow ovarian activities.

Subjects will have visits twice a week and sometimes more often to assess the effects of the pill on:

* cervical mucus properties by a cervical mucus sampling
* ovarian activity by a vaginal ultrasound (TVUS)
* reproductive hormones levels by a blood sample (Progesterone (P4), Estradiol (E2), Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH))
* plasma drug level by a blood sample

ELIGIBILITY:
Inclusion Criteria:

* Women in good overall health with no chronic medical conditions that result in periodic exacerbations that require significant medical care
* Women between 18 and 35 years inclusive at the screening visit
* BMI< 32 kg/m²
* Regular menstrual cycles between 21 and 35 days when not using hormonal contraception.

  * Subjects postpartum or post-abortal must have one normal menstrual cycle (2 menses) prior to enrollment.
  * Subjects previously using Intra-Uterine Device (IUD) or taking hormonal contraception (or any other hormonal treatment, except an injectable treatment) need to have at least one menstrual cycle (2 menses) without the treatment before screening.
  * Subject previously using an injectable (DMPA), must have had their last injection at least 9 months before screening.
* Women not at risk of pregnancy: not sexually active, or willing to protect all acts of intercourse with condoms, or have a sterile partner or have undergone previous tubal ligation (including validated Essure), or be in a same sex relationship.
* Women able to give informed consent form to participate in the study and in the opinion of the investigator able to follow all study requirements, use the study medication and record the requested information appropriately
* Intact uterus and both ovaries
* At least one progesterone concentration > 3 ng/mL (>10 nmol/L) during the luteal phase of the screening period

Exclusion Criteria:

* Pregnant as confirmed by positive high-sensitivity urine pregnancy test at enrollment visit
* Trying to conceive or desire to conceive in the next 3 months
* Currently breastfeeding, or within the last 2 months
* Known Polycystic Ovarian Syndrome (PCOS)
* Cancer (or past history of any carcinoma or sarcoma)
* Known abnormal thyroid status, if in clinical judgment of the investigator it cannot be controlled during the study
* Known hypersensitivity to the ingredients of the test active substances or its excipients
* Current acute liver disease and/or benign liver tumors
* Have vaginal or cervical infection including clinical evidence of bacterial vaginosis
* Evidence of abnormal cervical lesion
* History of excisional or ablative treatment procedure on cervix (ie. Loop Electrosurgical Excision Procedure (LEEP), Cryotherapy, Cold Knife Cone)
* Undiagnosed abnormal uterine bleeding
* Prior malabsorptive-type bariatric surgery
* Known or suspected alcoholism or illicit drug abuse
* Use of any hormonal contraception or IUD other than the study medication during the study (including ulipristal acetate for emergency contraception in the past 5 days)
* Use of any medications that can interfere with the metabolism of progestin-based contraceptives (e.g CYP3A4 enzymes inducers or inhibitors, etc)
* Unstable diabetes mellitus
* Current participation in any other trial of an investigational medicine or participation in the past two months (or within 5 elimination half-lives for chemical entities or 2 elimination half-lives for antibodies, whichever is the longer) before screening
* Abnormalities in laboratory results or TVUS performed at screening visit recognized as clinically significant by the investigator
* Conditions not suitable for frequent TVUS examinations, (e.g. virgo intacta)
* In custody or submitted to an institution due to a judicial order
* Relative or household member of the investigator's or sponsor's staff

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, MD, Principal Investigator — Oregon Health and Sciences University; Mitchell Creinin, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis, Sacramento, California
  - Oregon Health and Sciences University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edelman A, Hemon A, Creinin M, Borensztein P, Scherrer B, Glasier A. Assessing the Pregnancy Protective Impact of Scheduled Nonadherence to a Novel Progestin-Only Pill: Protocol for a Prospective, Multicenter, Randomized, Crossover Study. JMIR Res Protoc. 2021 Jun 8;10(6):e29208. doi: 10.2196/29208. PMID 33970869
- See also: World Health Organization Laboratory Manual for the Examination and Processing of Human Semen. Fifth edition 2010 — http://apps.who.int/iris/bitstream/handle/10665/44261/9789241547789_eng.pdf;jsessionid=9C2792C737959457E7FC8947BA13D21E?sequence=1://

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled subjects were randomized at the first visit of week 5 (first week of treatment period 2) in Arm A or B.
  All subjects received the same treatment during the first four weeks of treatment
Groups:
- Treatment Period 1: All Enrolled Subjects: Subjects were enrolled in treatment period 1 without being assigned an arm (Arm A or Arm B) until week 5.
  Subjects took norgestrel 75 mcg every day at the same time for three 28-day treatment periods, except for 1 specific day during treatment period 2 and treatment period 3
- Arm A: Delayed Then Missed Pill: Treatment period 2, visit Day 42+/- 3 days: 6 hour delayed intake of Norgestrel 75 mcg Treatment period 3, visit Day 70+/- 3 days: missed pill of Norgestrel 75 mcg
  Subjects took norgestrel 75 mcg every day at the same time for three 28-day treatment periods, except for 1 specific day during treatment period 2 and treatment period 3
- Arm B: Missed Then Delayed Pill: Treatment period 2, visit Day 42+/- 3 days: missed pill of Norgestrel 75 mcg Treatment period 3, visit Day 70+/-3 days: 6 hour delayed intake of the pill of Norgestrel 75 mcg
  Subjects took norgestrel 75 mcg every day at the same time for three 28-day treatment periods, except for 1 specific day during treatment period 2 and treatment period 3
Period: Treatment Period 1
Arm/Group | Treatment Period 1: All Enrolled Subjects | Arm A: Delayed Then Missed Pill | Arm B: Missed Then Delayed Pill
Started | 52 | 0 (Randomization in Treatment Period 2) | 0 (Randomization in Treatment Period 2)
Completed | 51 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Treatment Periods 2 and 3
Arm/Group | Treatment Period 1: All Enrolled Subjects | Arm A: Delayed Then Missed Pill | Arm B: Missed Then Delayed Pill
Started | 0 (Subjects having completed Treatment Period 1 randomized in Arm A or Arm B) | 26 | 25
Completed | 0 | 23 | 22
Not Completed | 0 | 3 | 3
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All subjects enrolled in the study
Groups:
- All Enrolled Subjects: All subjects enrolled in the study
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (4.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 38
  More than one race | 2
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 23.96 (3.65)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Delayed Intake or Missed Pill on Cervical Mucus Score (CMS)
Description: Difference in Cervical Mucus Score between baseline (as Day 41 or Day 69) and delayed (Day 42 and Day 70) or missed pill (Day 43 or day 71)
  The Insler cervical mucus score (0-12) is the sum of 4 subscores:
  * viscosity from 0 (thick, highly viscous) to 3 (watery,minimally viscous)
  * ferning from 0 (no crystallization) to 3 (tertiary and quaternary stem ferning)
  * spinnbarkeit from 0 (<1 cm) to 3 (>= 9 cm)
  * rank for cells from 0 (>20 cells per High Power Field or >1000 cells per μL) to 3 (0 cell)
  A score <5 is considered as a protective score while a score >9 is considered as a non protective score
Time Frame: Day 41 +/- 3 day to Day 43 +/3 days and Day 69 +/- 3 days to Day 71 +/-3 days
Population: Full Analysis Set for Primary endpoint: Subjects who had cervical mucus score for either D41-D43 or D69-71
Measure: Least Squares Mean (Standard Error); unit: changes in scores on a scale
Groups:
- Delayed Pill Intake: All the subjects of Arm A during treatment period 2 and all the subjects of Arm B during treatment period 3
  Norgestrel 0.075 mg: Subjects took norgestrel 75 mcg every day at the same time for three 28-day treatment periods, except for one specific day (Day 42 +/3 days) during treatment period 2 or treatment period 3 (Day 70 +/3 days) where they delayed their pill intake of 6 hours
- Missed Pill Intake: All the subjects of Arm B during treatment period 2 and all the subjects of Arm A during treatment period 3
  Norgestrel 0.075 mg: Subjects took norgestrel 75 mcg every day at the same time for three 28-day treatment periods, except for one specific day (Day 42 +/3 days) during treatment period 2 or treatment period 3 (Day 70 +/3 days) where they missed their pill
Arm/Group | Delayed Pill Intake | Missed Pill Intake
Number analyzed (Participants) | 46 | 47
changes in scores on a scale
  Difference in CMs after a 3-hour late pill: number analyzed (Participants) | 46 | 0
  Difference in CMs after a 3-hour late pill | 1.0 (0.3) |
  Difference in CMs after a 6-hour late pill: number analyzed (Participants) | 0 | 47
  Difference in CMs after a 6-hour late pill |  | 0.7 (0.3)
  Difference in CMs after a 24-hour late pill (missed pill): number analyzed (Participants) | 0 | 47
  Difference in CMs after a 24-hour late pill (missed pill) |  | 0.1 (0.3)
  Difference in CMS between 3h delay and next pill 18h later: number analyzed (Participants) | 46 | 0
  Difference in CMS between 3h delay and next pill 18h later | 0.3 (0.31) |
Statistical Analysis 1: Comparison: Delayed Pill Intake vs Missed Pill Intake; Mixed model for repeated measures using as response delta to Day41, delta to Day42, delta to Day70 and delta to Day71. Covariates: period, intervention (missed pill or delayed pill), sequence of intervention (missed pill then delayed pill and vice versa), time and subject. Subject as random effect + time repeated effect within each combination subject* period; Test type: Other — Is the overall mean change from baseline different from zero? Or did the infringement of schedule regardless the type of infringement lead to a change in mucus score?; p = 0.26, Mixed Models Analysis — P value from model testing intercept (does infringement change mucus score?) P-value from a repeated measures mixed model with the period, intervention, sequence and time (visit) as covariates. P-values ≤0.050 are considered significant

2. Secondary Outcome: Duration of Protective Effect of Cervical Mucus After a 6h Delayed or a Missed Pill
Description: Subjects are classified according to the risk of losing cervical mucus protection after a 6h delayed or a missed pill, on the day of the infringement and on the day after A cervical mucus score (CMS) <5 is considered as a protective score
  * Full protection: CMS stay <5 after both a delayed or a missed pill, on the day of infringement and on the day after.
  * Absence of risk increase: CMS stay <5 on the day of infringement and on the day after.
  * Transient risk increase: CMS increase >=5 on the day of infringement but go back to <5 on the day after.
  * Prolonged risk increase: CMS increase >=5 on the day of infringement and stay >=5 on the day after.
Time Frame: Day 41 +/- 3 day to Day 43 +/3 days and Day 69 +/- 3 days to Day 71 +/-3 days
Population: Full Analysis Set for Primary endpoint: Subjects who had cervical mucus score for either D41-D43 or D69-71 and a CMS at Baseline =< 5
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Pill Intake | Missed Pill Intake
Number analyzed (Participants) | 44 | 41
Participants
  Full Protection | 30 | 30
  Absence of risk increase | 38 | 37
  Transient risk increase | 5 | 4
  Prolonged risk increase | 1 | 0
Statistical Analysis 1: Comparison: Delayed Pill Intake vs Missed Pill Intake; Absence of risk increase; Test type: Other; p > 0.999, McNemar — p values > 0.050 (Not Statistically significant); McNemar test comparing agreement in the missed and delayed periods
Statistical Analysis 2: Comparison: Delayed Pill Intake vs Missed Pill Intake; Transient risk increase; Test type: Other; p = 0.655, McNemar — p values > 0.050 (Not Statistically significant); McNemar test comparing agreement in the missed and delayed periods
Statistical Analysis 3: Comparison: Delayed Pill Intake vs Missed Pill Intake; Prolonged risk increase; Test type: Other; p = 0.317, McNemar — p values > 0.050 (Not Statistically significant); McNemar test comparing agreement in the missed and delayed periods

3. Secondary Outcome: Ovarian Status (OS)
Description: Ovarian Status (OS) defined as:
  * OSq = quiescence defined as an Ovarian Activity Score (OAS) =< 3
  * OSa = active defined as OAS = 4 or 5
  * OSalp = ovulation with abnormal luteal phase defined as OAS = 6 at only one visit
  * OSnlp = ovulation with normal luteal phase as defined as OAS = 6 at two consecutive visits or OAS = 7
  Ovarian Activity Score between 1 and 7:
  * 1= No ovarian activity
  * 2= Potential activity
  * 3= Non-active follicle like structure
  * 4= Active follicle like structure
  * 5= Postovulatory, low progesterone level
  * 6= Postovulatory, intermediate progesterone level
  * 7= Postovulatory, high progesterone level
Time Frame: From Day 1 to Day 84 (if no follow-up) or up to Day 90 (if follow-up)
Population: Full Analysis Set - Ovarian Activity: Subjects with an Ovarian Status (OS) for either Treatment Period 2 or Treatment Period 3
Measure: Count of Participants; unit: Participants
Groups:
- OS: Reported Perfect Use Period (Treatment Period 1): Subjects in Treatment Period 1 who also had an Ovarian Status in either Treatment Period 2 or Treatment Period 3
- OS: Delayed Pill Period: Subjects with Ovarian Status, of:
  * Arm A in Treatment Period 2
  * Arm B in Treatment Period 3
- OS: Missed Pill Period: Subjects with Ovarian Status, of:
  * Arm A in Treatment Period 3
  * Arm B in Treatment Period 2
Arm/Group | OS: Reported Perfect Use Period (Treatment Period 1) | OS: Delayed Pill Period | OS: Missed Pill Period
Number analyzed (Participants) | 49 | 46 | 46
Participants
  OSq | 7 | 10 | 7
  OSa | 25 | 22 | 25
  OSalp | 5 | 4 | 2
  OSnlp | 12 | 10 | 12
Statistical Analysis 1: Comparison: OS: Reported Perfect Use Period (Treatment Period 1) vs OS: Delayed Pill Period; A stratified McNemar test (stratification on the site, AGREE option in SAS) was used to compare the distribution of ovarian activity classification in the perfect use period to the delayed and missed pill periods (pairwise vs perfect use). The worst (meaning most risk of ovulation) ovarian activity category in the period was used for the analyses; Test type: Other; p < 0.001, McNemar — Indicates significance at the 0.05 level (p-value ≤ 0.05); P-value from an exact kappa test comparing agreement of ovarian status vs the reported perfect use period
Statistical Analysis 2: Comparison: OS: Reported Perfect Use Period (Treatment Period 1) vs OS: Missed Pill Period; [analysis description as in outcome 3, analysis 1]; Test type: Other; p < 0.001, McNemar — Indicates significance at the 0.05 level (p-value ≤ 0.05); P-value from an exact kappa test comparing agreement of ovarian status vs the reported perfect use period

4. Secondary Outcome: Cervical Mucus Protection
Description: Higher Cervical Mucus Score (CMS) in:
  * Treatment Period 1 (Reported Perfect Use Period)
  * Delayed pill period: Treatment Period 2 for Arm A and Treatment Period 3 for Arm B
  * Missed pill period: Treatment Period 3 for Arm A and Treatment Period 2 for Arm B
  A score =< 4 is considered as a protective score and a score >= 9 is considered as a non protective score
Time Frame: From Day 1 to Day 84
Population: Full Analysis Set - Mucus Secondary: Subjects who had cervical mucus scores for at least 7 visits for either Treatment Period 2 or Treatment Period 3
Measure: Count of Participants; unit: Participants
Groups:
- CMS: Reported Perfect Use Period (Treatment Period 1): Subjects in Treatment Period 1 who had at least 7 cervical mucus scores in either Treatment Period 2 or Treatment Period 3
- CMS: Delayed Pill Period: Subjects who had at least 7 cervical mucus scores in:
  * Arm A: Treatment Period 2
  * Arm B: Treatment Period 3
- CMS: Missed Pill Period: Subjects who had at least 7 cervical mucus scores in:
  * Arm A: Treatment Period 3
  * Arm B: Treatment Period 2
Arm/Group | CMS: Reported Perfect Use Period (Treatment Period 1) | CMS: Delayed Pill Period | CMS: Missed Pill Period
Number analyzed (Participants) | 49 | 47 | 47
Participants
  CMS <=4 | 32 | 27 | 28
  CMS between 5 & 8 (inclusive) | 17 | 20 | 15
  CMS >=9 | 0 | 0 | 4
Statistical Analysis 1: Comparison: CMS: Reported Perfect Use Period (Treatment Period 1) vs CMS: Delayed Pill Period; Stratified McNemar test (stratification on the site, AGREE option in SAS) to compare the distribution of cervical mucus scores in the perfect use period to the delayed and missed pill periods (pairwise vs perfect use); Test type: Other; p = 0.127, McNemar; P-value from an exact kappa test comparing agreement of cervical mucus score classification vs the reported perfect use period
Statistical Analysis 2: Comparison: CMS: Reported Perfect Use Period (Treatment Period 1) vs CMS: Missed Pill Period; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.018, McNemar — * Indicates significance at the 0.05 level (p-value ≤ 0.05); [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Conception Protection Risk
Description: Binary analysis of whether a subject is at risk of conception based only on their ovarian status (OS) and cervical mucus score (CMS) the days before ovulation:
  Are considered protected, subjects with OSq, OSa OR CMS =<4 Are considered at risk, subjects with OSalp or OSnlp AND CMS >=5
Time Frame: Day 1 to Day 84 (up to Day 90 if follow-up)
Population: Full Analysis Set - Conception: Subjects who had a OS + enough CMS to assess their Conception Protection Risk & Level in either Treatment Period 2 or Treatment Period 3
Measure: Count of Participants; unit: Participants
Groups:
- CP/R&L: Reported Perfect Use Period (Treatment Period 1): Subjects in Treatment Period 1 who had a OS + enough CMS to assess their Conception Protection Risk & Level in either Treatment Period 2 or Treatment Period 3
- CP/R&L: Delayed Pill Period: Subjects who had a OS + enough CMS to asses their Conception Protection Risk & Level in:
  * Arm A: Treatment Period 2
  * Arm B: Treatment Period 3
- CP/R&L: Missed Pill Period: Subjects who had a OS + enough CMS to assess their Conception Protection Risk & Level in:
  * Arm A: Treatment Period 3
  * Arm B: Treatment Period 2
Arm/Group | CP/R&L: Reported Perfect Use Period (Treatment Period 1) | CP/R&L: Delayed Pill Period | CP/R&L: Missed Pill Period
Number analyzed (Participants) | 49 | 46 | 46
Participants
  Protected | 46 | 42 | 41
  At risk | 3 | 4 | 5

6. Secondary Outcome: Conception Protection Level
Description: Ternary analysis of the level of protection from conception of subjects, based only on the ovarian status (OS) and cervical mucus score (CMS) the days before ovulation:
  * Minimum protection or unlikely to be protected: OSnlp and CMS ≥ 9
  * Medium protection or likely to be protected: OSnlp and CMS comprised between 5 and 8 or OSalp and CMS ≥ 5
  * Maximum protection or highly likely to be protected: OSq or OSa or a CMS ≤ 4
Time Frame: Day 1 to Day 84 (up to Day 90 if follow-up)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | CP/R&L: Reported Perfect Use Period (Treatment Period 1) | CP/R&L: Delayed Pill Period | CP/R&L: Missed Pill Period
Number analyzed (Participants) | 49 | 46 | 46
Participants
  Maximum/Highly Likely to be Protected | 46 | 42 | 41
  Medium/Likely to be Protected | 3 | 4 | 3
  Minimum/Unlikely to be Protected | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: From Day 1 to Day 84
Description: Systematic Assesment:
  * Adverse Events collected at each visit
  * Hematology, Chemistry, Vital Signs collected at End of Study visit
  * Vaginal Bleedings recorded daily by subjects in a diary
Groups:
- All Enrolled Subjects: All subjects enrolled in the study.
  The adverse events were reported for all the subjects enrolled in the study for the entire length of the study.
  The subjects were randomized in their respective arm in week 5. Subjects in Arm A had a 6 hour delayed pill at Day 42 +/- 3 days and a missed pill at Day 70+/- 3 days while subjects in Arm B had a missed pill at Day 70+/- 3 days and a 6 hour delayed pill at Day 42 +/- 3 days.
  It was considered that the difference in investigational medication intake between the arms would not have an impact on adverse event's frequency, so the adverse events were reported for all subjects enrolled, whatever the arm they were assigned to, and for the entire length of the study.
- Perfect Use Period: All the subjects having starting treatment period 1.
  Affected participants by an adverse event during this treatment period are reported out of the total of subjects having started the treatment period 1.
- Delayed Pill Intake: Subjects having started a delayed pill period, meaning treatment period 2 for subjects randomized in week 5 in Arm A, and treatment period 3 for subjects in Arm B
  Affected participants by an adverse event during this treatment period are reported out of the total of subjects having started this treatment period.
- Missed Pill Intake: Subjects having started a missed pill period, meaning treatment period 3 for subjects randomized in week 5 in Arm A, and treatment period 2 for subjects in Arm B
  Affected participants by an adverse event during this treatment period are reported out of the total of subjects having started this treatment period.
Arm/Group | All Enrolled Subjects | Perfect Use Period | Delayed Pill Intake | Missed Pill Intake
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52 | 0/50 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/52 | 1/50 | 0/48
Other Adverse Events (participants affected / at risk) | 50/52 | 42/52 | 29/50 | 33/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=52) | Perfect Use Period (N=52) | Delayed Pill Intake (N=50) | Missed Pill Intake (N=48)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Anaphylaxis Reaction with difficulty breathing. Severe. Recovered/Resolved Not Related to study medication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Enrolled Subjects (N=52) | Perfect Use Period (N=52) | Delayed Pill Intake (N=50) | Missed Pill Intake (N=48)
Metrorrhagia (Reproductive system and breast disorders) | 41 | 23 | 13 | 15
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 16 | 6 | 7 | 6
Acne (Skin and subcutaneous tissue disorders) | 11 | 9 | 0 | 2
Breast tenderness (Reproductive system and breast disorders) | 6 | 5 | 1 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 5 | 1 | 2 | 2
Fatigue (General disorders) | 5 | 4 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 5 | 1 | 2 | 2
Vulvovaginal discomfort (Reproductive system and breast disorders) | 5 | 0 | 2 | 3
Headache (Nervous system disorders) | 4 | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 1 | 1
Muscle spams (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 3 | 2 | 1 | 0
Uterine spasm (Reproductive system and breast disorders) | 3 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT03585712/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT03585712/SAP_001.pdf